CLINICAL TRIAL: NCT02696200
Title: Novel Protection Against Potential Brain Injury During Competitive Football Head Impacts
Brief Title: Protection Against Potential Brain Injury During Competitive Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-2205
Record Dates: First submitted 2015-05-28; First posted 2016-03-02 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects Wearing the Q Collar (Experimental): Subjects wearing the Q collar throughout the football season
  Interventions: Device: Q Collar
- Subjects Not Wearing the Q Collar (No Intervention): Control group of subjects not wearing the q collar

INTERVENTIONS:
Device: Q Collar — The device is fitted to the neck to provide a comfortable and precise jugular compression that potentially mitigates cerebral slosh. The device will be worn inside the collar of an athletic compression shirt.
  Arms: Subjects Wearing the Q Collar

SUMMARY:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver (the Device). Preliminary research suggests that the Device has the potential to reduce the likelihood of TBI. The currently developed collar has been approved for studies in humans and the results indicate safety for use during high demand and maximal exertion activities, This study will investigate the effectiveness of this device in high school athletes playing a collision sport such as football. The use of helmets during such a high-risk sport will allow for collision measurement devices to be embedded in the helmet and will not affect play or fit of equipment. Athletes participating in this study will be randomly assigned to one of two groups: 1) Device wearing during the season or 2) Non-device wearing during the season. The helmets of all participants will be outfitted with an accelerometer which will measure the magnitude of every impact to the head sustained by the athlete. Effectiveness of the device will be determined via differences in longitudinal brain imaging and functional testing following competitive football participation. A subset of athletes who report a diagnosed concussion will also receive additional brain neuroanatomical and neurophysiological testing within a week following the diagnosed concussive event. The purpose of the study is to monitor longitudinal changes in brain structure and function between the preseason and postseason, in a population of football playing athletes wearing the Device and compared to a similar population not wearing the device. Secondly, the purpose is to determine the protection of the device relative to amount and magnitude of sustained head impacts.

DETAILED DESCRIPTION:
The Device has the promise of providing a novel mechanism for reducing or preventing the likelihood of TBI, and may be used in conjunction with other protective equipment. TBI is the leading cause of death in individuals under age 45. The cost of TBI in the U.S. is estimated at anywhere from $50 to $150 billion, annually. The January, 2008 New England Journal of Medicine reports, "Head and neck injuries, including severe brain trauma, have been reported in one quarter of service members who have been evacuated from Iraq and Afghanistan". The vast majority of these injuries have resulted from exposure to improvised explosive device (IED) blast waves. Head injuries, concussions and the resulting trauma have been in public discussion recently as the National Football League (NFL) deals with a lawsuit regarding head injuries by about one-third of living former NFL players.

According to NASA, "The oscillation of a fluid caused by an external force, called sloshing, occurs in moving vehicles containing liquid masses, such as trucks, etc." This oscillation occurs when a vessel is only partially filled. It is hypothesized that the brain faces similar slosh energy absorption during external force impartation. Slosh permits external energies to be absorbed by the contents of a partially filled vessel or container by means of inelastic collisions. Tissues of differing densities can decelerate at different rates creating shear and cavitation. If the collisions between objects or molecules are elastic, the transfer of energies to those objects diminishes, minimizing the energies imparted by slosh.

Woodpeckers, head ramming sheep and all mammals (including humans) have small, little known and misunderstood muscles in their necks called the omohyoid muscles. Highly G-tolerant creatures of the forest have utilized these muscles to gently restrict outflow of the internal jugular veins thereby "taking up" the excess compliance of the cranial space and ultimately protecting themselves from TBI like tiny "airbags" in a motor vehicle. Rat studies by have demonstrated that we can easily and safely facilitate this muscle's actions by a well-engineered gentle compression over those muscles.

The medical Queckenstedt Maneuver devised to detect spinal cord compression, gently places pressure over the external jugular veins to increase cerebral spinal volume and pressure. In this maneuver, the veins are compressed while a lumbar puncture monitors the intracranial pressure. "Normally, the pressure rise to the higher 'plateau' level occurs instantly upon jugular compression to fall again equally fast upon release of the compression". This incredibly simple principle can be employed to protect soldiers and athletes from TBI by safely, and reversibly, increasing intracranial volume and pressure. The neck collar device is made of Outer collar - hytrel (thermoplastic elastomer), Inner collar - TPSiV (thermoplastic elastomer), metal insert (stainless steel), and is fitted to the neck to provide a comfortable and precise jugular compression that potentially mitigates cerebral slosh.

Although the skull, blood, and brain are "almost incompressible," the vasculature tree of the cerebrum is quite reactive and compressible. As volume is added to the cranium, eventually the compensatory reserve volume is surpassed and the intracranial pressure increases slightly. Increasing cerebral blood volume by just 1-3% safely and reversibly reduces compliance of the cerebral vascular tree and diminishes absorption of slosh energies. Jugular compression increases cerebral blood volume almost instantaneously. As mentioned, this degree of increase has significantly mitigated slosh and TBI in laboratory animals and mimics the highly concussion resistant wild animals that are able to reflexively increase cerebral blood volume through natural jugular compression.

A landmark article, published in the Journal of Neurosurgery, used a standard acceleration-deceleration impact laboratory model of mild TBI. The study showed a successful and marked reduction of axonal injury following Internal Jugular Vein (IJV) compression as indicated by immunohistochemical staining of Amyloid Precursor Proteins (APP). It is argued that IJV compression reduces slosh-mediated brain injury by increasing intracranial blood volume and reducing the compliance and potential for brain movement within the confines of the skull. The potential for such technique to mitigate both linear and rotational brain injury in humans by "internal protection" represents the most novel approach to mitigating TBI.

The current project will be designed following a prospective longitudinal study design. All MRI scanning will be performed on a 3 Tesla Philips Achieva MRI scanner located in Imaging Research Center (IRC) in the Cincinnati Children's Hospital Research Foundation (CCHRF). Sedation will not be used for any of the test visits. The entire MRI series, including anatomical imaging, DTI, resting state fMRI, SWI, HARDI, ASL and BOLD will be completed in 65 minutes or less (see Table 1 for detailed specifications). All functional and neurocognitive testing will be performed at the Cincinnati Children's Hospital Human Performance Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent
* Must be 14 years or older and a participant on varsity level high school football team

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinanti Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published however individual participant data will remain secure.

REFERENCES:
- [Derived] Yuan W, Leach J, Maloney T, Altaye M, Smith D, Gubanich PJ, Barber Foss KD, Thomas S, DiCesare CA, Kiefer AW, Myer GD. Neck Collar with Mild Jugular Vein Compression Ameliorates Brain Activation Changes during a Working Memory Task after a Season of High School Football. J Neurotrauma. 2017 Aug 15;34(16):2432-2444. doi: 10.1089/neu.2016.4834. Epub 2017 Jun 8. PMID 28437225
- [Derived] Myer GD, Yuan W, Barber Foss KD, Thomas S, Smith D, Leach J, Kiefer AW, Dicesare C, Adams J, Gubanich PJ, Kitchen K, Schneider DK, Braswell D, Krueger D, Altaye M. Analysis of head impact exposure and brain microstructure response in a season-long application of a jugular vein compression collar: a prospective, neuroimaging investigation in American football. Br J Sports Med. 2016 Oct;50(20):1276-1285. doi: 10.1136/bjsports-2016-096134. Epub 2016 Jun 15. PMID 27307271

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar
Started | 32 | 30
Completed | 32 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 30 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Determine Average Number of Hits Between Groups
Description: monitor the differences in average number of hits between the group wearing the collar and the group not wearing the collar
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: number of hits
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar
Number analyzed (Participants) | 32 | 30
number of hits
  Avg # of hits >20g | 896.43 (600.03) | 795.40 (508.92)
  Avg # of hits >50g | 144.67 (106.55) | 145.85 (109.98)
  Avg # of hits >100g | 14.38 (11.29) | 18.3 (20.85)
  Avg # of hits >150g | 2.43 (3.11) | 1.8 (2.04)
  Avg # of hits >200g | 0.43 (1.17) | 0.30 (0.73)

2. Primary Outcome: Number of Participants Undergoing EEG Assessment
Description: determine the number of subjects in the collar group and the non collar group that underwent EEG assessment
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar
Number analyzed (Participants) | 32 | 30
Participants | 32 | 30

3. Primary Outcome: Change in Fractional Anisotropy (FA)
Description: Change in fractional anisotropy (FA) from Pre to Post season
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar
Number analyzed (Participants) | 32 | 30
percentage of change | 0.03 (1.24) | 2.43 (1.01)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Subjects Wearing the Q Collar | Subjects Not Wearing the Q Collar
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02696200/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT02696200/Prot_SAP_001.pdf